CLINICAL TRIAL: NCT03256435
Title: PrEP Uptake, Adherence, and Retention for African American MSM in Mississippi
Brief Title: Retention in PrEP Care for African American MSM in Mississippi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Mississippi Medical Center (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1611001642; 5R34MH109371-03 (NIH)
Record Dates: First submitted 2017-04-14; First posted 2017-08-22 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Preventive Medicine; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): RAMP PrEP initiation, adherence, and retention intervention package as well as standard of care (access to a financial advocate and clinical staff to support, facilitate, and assist in linkage to the established PrEP clinic at Open Arms and to facilitate initiation of, and obtaining, PrEP medications)
  Interventions: Behavioral: RAMP PrEP initiation, adherence, and retention intervention
- Control Arm (No Intervention): Standard of care (access to a financial advocate and clinical staff to support, facilitate, and assist in linkage to the established PrEP clinic at Open Arms and to facilitate initiation of, and obtaining, PrEP medications)

INTERVENTIONS:
Behavioral: RAMP PrEP initiation, adherence, and retention intervention — The intervention arm will receive facilitated strengths-based case management (SBCM)-delivered by trained interventionists-to help navigate the PrEP medical care system and support the participant and health care staff in meeting the challenges faced with obtaining PrEP medication (e.g., overcoming insurance barriers or barriers with co-pays). This also includes facilitated integration into the PrEP clinic and obtaining monthly PrEP prescription refills.
  Arms: Treatment Arm

SUMMARY:
Innovative and novel HIV prevention interventions are urgently needed for African American (AA) young men who have sex with men (YMSM) in the South, and in Mississippi in particular. HIV pre-exposure prophylaxis (PrEP) is a newer HIV prevention strategy that consists of a daily oral antiretroviral pill taken on an ongoing basis by HIV-uninfected but at-risk individuals. Although acceptability studies have demonstrated high interested in PrEP in the US, uptake remains limited. To date, studies of PrEP initiation have largely been limited to settings in which PrEP is provided free of charge. Barriers to PrEP initiation and retention in PrEP care in real world settings are likely more complex, since payment for PrEP can be a substantial financial burden.

The ADAPT_ITT approach (an approach to adapting behavioral interventions to new populations: Assessment, Decision, Administration, Production, Topical Experts - Integration, Training, Testing) will be used to develop and pilot test a RAMP (Retain African American Men in PrEP) intervention that aims to promote PrEP adherence and retention in care in Jackson, MS and focuses on recruiting AA YMSM in a city with some of the highest HIV infection rates in the country. This study will include formative research to understand the cultural and social contexts that influence AA YMSM's PrEP use patterns and the acceptability of our proposed intervention. Results from these qualitative interviews will inform the study intervention which will be tested and refined in a dynamic open pilot evaluation.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) bear a disproportionate burden of the HIV epidemic in the United States (US), and the number of new HIV diagnoses among MSM is increasing every year. Despite HIV incidence remaining relatively stable overall, HIV incidence is increasing among MSM, and among Black/African American (hereafter AA) young MSM (YMSM) in particular. Black/AA MSM represent less than 1% of the population but account for 25% of new HIV diagnoses. Compared to MSM of other races, AA MSM are 3 times more likely to be HIV infected. Among YMSM, the disparities are greatest; AA MSM aged 20-29 have an HIV prevalence of 34%, whereas White MSM in the same age range have an HIV prevalence of 5.5%. Additionally, the American South accounts for 46% of new HIV diagnoses in the US and 45% of new AIDS diagnoses. Mississippi is ranked 7th in the country in HIV case rates, with an overall rate of 20.7 per 100,000 persons; however, some census tracts have rates of 2-5%, which is comparable to some sub-Saharan African countries. There are alarming racial disparities related to HIV/AIDS; in Mississippi, AAs comprise 37% of the population but accounted for 76% of HIV infection reported in 2013. Between 2011 and 2013, the number of infections among MSM in Mississippi increased 43%, with an even sharper increase among AA YMSM, who have among the highest rates of infection in the nation.

Given the disproportionate burden of HIV, worse HIV outcomes, and current social climate, innovative and novel HIV prevention interventions are urgently needed for AA YMSM in the South, and in Mississippi in particular. HIV pre-exposure prophylaxis (PrEP) is a newer HIV prevention strategy that consists of a daily oral antiretroviral pill taken on an ongoing basis by HIV-uninfected but at-risk individuals. Its efficacy has been well established in randomized controlled trials and open-label studies for MSM and other groups. Although acceptability studies have demonstrated high interest in PrEP in the US, uptake remains limited. To date, studies of PrEP initiation have largely been limited to settings in which PrEP is provided free of charge. Barriers to PrEP initiation and retention in PrEP care in real world settings are likely more complex, since payment for PrEP can be a substantial financial burden. Although most health insurance programs are covering the cost of PrEP, and the industry-sponsored PrEP Medication Assistance Program exists to assist people who do not have insurance, these programs require patient and clinician awareness, sufficient staffing and appropriate infrastructure.

A body of evidence is only beginning to emerge related to PrEP adherence and little is known about retention in PrEP care, most of which is in the context of either RCTs or open-label studies in which PrEP is provided free of charge. The efficacy of PrEP is closely tied to adherence, and evidence suggests that efficacy decreases exponentially with fewer doses of PrEP per week; maximum efficacy is achieved when 6-7 doses are taken per week, but PrEP provides high protection with at least 4 doses per week. In an open label study of PrEP uptake and adherence in MSM, 71% of participants receiving PrEP had drug detected after initiation of PrEP. AA YMSM in Jackson, MS face many challenges to optimal adherence and retention in care, including inconsistent routines, socioeconomic challenges, and logistical difficulty in returning for follow-up visits. MSM may not want to disclose use of PrEP to family or friends, due to the potential for unintended disclosure of sexual orientation, which may result in reduced social support for PrEP adherence or returning for care. Understanding barriers and facilitators to adherence and retention in care for AA YMSM, and subsequently the development of interventions to improve them, will be necessary to ensure maximum PrEP effectiveness.

The ADAPT_ITT approach will be used to develop and pilot test a RAMP intervention that aims to promote PrEP adherence and retention in care in Jackson, MS and focuses on recruiting AA YMSM in a city with some of the highest HIV infection rates in the country. This study will include formative research to understand the cultural and social contexts that influence AA YMSM's PrEP use patterns and the acceptability of our proposed intervention. Results from these qualitative interviews will inform the study intervention which will be tested and refined in a dynamic open pilot evaluation.

Qualitative interviews (Phase 1) will "assess" individual, interpersonal and structural contexts of sexual risk behavior, anticipated adoption and use of new prevention technologies, barriers and facilitators to PrEP initiation and adherence, and optimal content and format for a PrEP initiation and adherence intervention. Using results of the qualitative interviews and input from key opinion leaders, the investigators will "decide" on intervention components and structure of the intervention package. The investigators will then "adapt" the Life-Steps intervention to be responsive to the unique context and complex needs of AA YMSM in Jackson, and "produce" a draft of the intervention manual. Our study team is made up of "topical experts" who will all have a central role in developing the intervention manual. Moreover, the open pilot evaluation (Phase 2) will be used to obtain further input on the draft intervention manual and protocol. After "integrating" the feedback obtained from the open pilot evaluation and exit interviews into the intervention manual and protocol, study staff will be "trained" in all final study procedures, and a provisional theory-based intervention to overcome barriers to PrEP adherence and retention, and reduce sexual risk behavior, among AA YMSM will be "tested" in a pilot Randomized Control Trial (RCT) (Phase 3). This intervention will have broad generalizability for AA YMSM across the South and the country as PrEP programs expand nationwide.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* assigned male sex at birth
* African American race
* report having sex with another person assigned male at birth who identifies as a man within the last year
* report behavioral risk for HIV infection (consistent with the CDC guidelines for prescribing PrEP: unprotected anal intercourse (UAI) with at least one HIV-infected or unknown serostatus partner in the preceding 6 months)
* HIV-uninfected by antibody test
* able to understand and speak English (for consenting and counseling).

Exclusion Criteria:

* unable to provide informed consent, including people with severe mental illness requiring immediate treatment or with mental illness limiting their ability to participate
* for aims 2 and 3 only, participants who are positive for Hepatitis B antigen or diagnosed with renal insufficiency (Glomerular Filtration Rate<50)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Presence of PrEP drug in blood samples | measured at 3 months
  Blood samples will be collected from participants at 3- and 6-month assessments to test for the presence of detectable levels of Emtricitabine/Tenofovir (FTC/TDF). Samples will be processed and shipped to Dr. Peter Anderson's lab at the University of Colorado Anschutz for analysis of the quantification (drug levels) of detectable serum levels of FTC and TDF.
Presence of PrEP drug in blood samples | measured at 6 months
  Blood samples will be collected from participants at 3- and 6-month assessments to test for the presence of detectable levels of Emtricitabine/Tenofovir (FTC/TDF). Samples will be processed and shipped to Dr. Peter Anderson's lab at the University of Colorado Anschutz for analysis of the quantification (drug levels) of detectable serum levels of FTC and TDF.
Self-reported adherence | measured at 3 months
  Self-reported adherence (with interviews) will supplement biological monitoring data at 3-month intervals, as well at the time of the intervention sessions (for both those in the intervention and comparison condition)
Self-reported adherence | measured at 6 months
  Self-reported adherence (with interviews) will supplement biological monitoring data at 3-month intervals, as well at the time of the intervention sessions (for both those in the intervention and comparison condition)

SECONDARY OUTCOMES:
PrEP Retention in Care over time | measured at 3 months
  This study will employ the Center for Disease Control (CDC) guidelines for retention in PrEP care, which include PrEP clinical visits every 3 to 6 months. "Retention in care" is defined as two PrEP follow up visits by month 8 of enrollment. While participants will only be randomized after attending the first PrEP clinic visit and receive a prescription from the study clinician for FTC/TDF, it is possible that they will not fill the prescription. The investigators will obtain a medical release from the participants in order that, at each assessment time-point, the study clinician can follow up with the pharmacy to determine whether or not the prescription was filled and picked up, and the date it was picked up (to assess time to initiation). Moreover, attendance at follow up clinic visits (months 3 and 6) will be calculated to assess retention in PrEP clinical care.
PrEP Retention in Care over time | measured at 6 months
  This study will employ the Center for Disease Control (CDC) guidelines for retention in PrEP care, which include PrEP clinical visits every 3 to 6 months. "Retention in care" is defined as two PrEP follow up visits by month 8 of enrollment. While participants will only be randomized after attending the first PrEP clinic visit and receive a prescription from the study clinician for FTC/TDF, it is possible that they will not fill the prescription. The investigators will obtain a medical release from the participants in order that, at each assessment time-point, the study clinician can follow up with the pharmacy to determine whether or not the prescription was filled and picked up, and the date it was picked up (to assess time to initiation). Moreover, attendance at follow up clinic visits (months 3 and 6) will be calculated to assess retention in PrEP clinical care.
Sexual risk behavior/behavioral adjustment | measured at baseline
  This study will use the AIDS-Risk Behavior Assessment (ARBA), a validated computerized self-interview designed to assess self-reported sexual behaviors. Sexual risk questions refer to 3 types of sexual behavior (anal, oral, vaginal) and assess detailed partner-by-partner sexual risk information by partner type (transactional, casual, main) and by HIV-status, protected/unprotected sex, and whether in the context of substance use in the prior 3 months.
Sexual risk behavior/behavioral adjustment | measured at 3 months
  This study will use the AIDS-Risk Behavior Assessment (ARBA), a validated computerized self-interview designed to assess self-reported sexual behaviors. Sexual risk questions refer to 3 types of sexual behavior (anal, oral, vaginal) and assess detailed partner-by-partner sexual risk information by partner type (transactional, casual, main) and by HIV-status, protected/unprotected sex, and whether in the context of substance use in the prior 3 months.
Sexual risk behavior/behavioral adjustment | measured at 6 months
  This study will use the AIDS-Risk Behavior Assessment (ARBA), a validated computerized self-interview designed to assess self-reported sexual behaviors. Sexual risk questions refer to 3 types of sexual behavior (anal, oral, vaginal) and assess detailed partner-by-partner sexual risk information by partner type (transactional, casual, main) and by HIV-status, protected/unprotected sex, and whether in the context of substance use in the prior 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Nunn, ScD, Principal Investigator — Brown University
Locations (1):
- Open Arms Clinic, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goedel WC, Coats CS, Chan PA, Sims-Gomillia CE, Brock JB, Ward LM, Mena LA, Nunn AS. A Pilot Study of a Patient Navigation Intervention to Improve HIV Pre-exposure Prophylaxis Persistence Among Black/African American Men Who Have Sex With Men. J Acquir Immune Defic Syndr. 2022 Jul 1;90(3):276-282. doi: 10.1097/QAI.0000000000002954. PMID 35312652